CLINICAL TRIAL: NCT02221063
Title: Thiamin Fortified Fish Sauce as a Means of Combating Infantile Beriberi in Rural Cambodia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Helen Keller International (Other); Grand Challenges Canada (Other); International Development Research Centre, Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: H14-00103; S6 0490-01-10 (Other: Grand Challenges Canada)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Thiamin Deficiency
Keywords: thiamin; thiamin diphosphate; beriberi; Cambodia; fish sauce; fortification; pregnancy; breastfeeding; childbearing age
MeSH Terms: conditions — Beriberi; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- low [thiamin] fortified fish sauce (Active Comparator): Fish sauce will contain 2 mg thiamin hydrochloride / mL fish sauce + iron (as NaFeEDTA)
  Interventions: Other: Thiamin fortified fish sauce (low concentration)
- higher [thiamin] fortified fish sauce (Active Comparator): Fish sauce will contain 8 mg thiamin hydrochloride / mL fish sauce + iron (as NaFeEDTA)
  Interventions: Other: Thiamin fortified fish sauce (higher concentration)
- Placebo fish sauce (Placebo Comparator): Fish sauce will contain only iron (as NaFeEDTA), no thiamin
  Interventions: Other: Placebo fish sauce

INTERVENTIONS:
Other: Thiamin fortified fish sauce (low concentration) — Low concentration thiamin fortified fish sauce will be consumed ad libitum for 6 months, with biweekly monitoring and evaluation to assess fish sauce usage by household and to re-stock fish sauce within the home.
  Arms: low [thiamin] fortified fish sauce
Other: Thiamin fortified fish sauce (higher concentration) — Higher concentration thiamin fortified fish sauce will be consumed ad libitum for 6 months, with biweekly monitoring and evaluation to assess fish sauce usage by household and to re-stock fish sauce within the home.
  Arms: higher [thiamin] fortified fish sauce
Other: Placebo fish sauce — Fish sauce fortified only with iron, not thiamin, will be consumed ad libitum for 6 months, with biweekly monitoring and evaluation to assess fish sauce usage by household and to re-stock fish sauce within the home.
  Arms: Placebo fish sauce

SUMMARY:
The purpose of this study is to determine whether consumption of thiamin fortified fish sauce over 6 months increases the thiamin status of women to a level consistent with a low risk of infantile beriberi. The investigators hypothesize that consumption of thiamin-fortified fish sauce will increase red blood cell thiamin concentrations, an indicator of thiamin status, in women consuming thiamin-fortified fish sauce, while concentrations will not change in women consuming a placebo fish sauce that does not contain thiamin.

DETAILED DESCRIPTION:
Purpose The purpose of this three-armed, double blind randomized control trial is to determine whether thiamin-fortified fish sauce is an efficacious means of increasing dietary thiamin intake in Cambodian women to a level that increases erythrocyte thiamin diphosphate (TDP) concentrations to a level consistent with a low risk of infantile beriberi. Two groups of women will participate in this study: women of childbearing age (18-45y; n=270), and pregnant women (18-45y; ~26 weeks pregnant at baseline; n=90).

Hypothesis Intervention with thiamin-fortified fish sauce will increase women's TDP concentrations to levels consistent with a low risk of infantile beriberi compared to those receiving the control fish sauce.

Study Justification Beriberi is a micronutrient deficiency disease caused by a lack of thiamin (vitamin B1) in the diet. Infantile beriberi is common in Southeast Asia.

Beriberi, a disease caused by severe thiamin deficiency, is rare in the west but is thought to be more common in developing countries, particularly those in Southeast Asia. In infants, beriberi presents with symptoms of heart failure and is fatal unless thiamin treatment is initiated immediately. Beriberi typically presents in exclusively breastfed infants whose mothers have suboptimal thiamin status and consequently have low breast milk thiamin concentrations. Maternal thiamin deficiency in Cambodia is likely a result of multiple factors: the high consumption of white, polished rice, which has been removed from its B-vitamin-containing husk, a lack of parboiling rice, and low dietary diversity. Improving the thiamin status of pregnant and lactating women is essential for combating infantile beriberi. Fortification of a food staple has proven to be a successful strategy in increasing population levels of thiamin because as a 'passive' intervention, it requires little to no behavior change. Fish sauce is an ideal vehicle for thiamin fortification: it is consumed daily in consistently high quantities, and is produced in centralized plants, and has been successfully used in Cambodia and Vietnam as a vehicle for iron fortification.

Research Method All villages in Prey Veng province that are not already involved in an active intervention (for example, homestead food production, micronutrient powder intervention etc) will be randomized. A Khmer-speaking research assistant will contact the Village Chief and/or Village Health Volunteer in the first village on the randomized list and determine the number of eligible women of childbearing age and pregnant women (~26 weeks) in that village. The research assistant will move down the randomized list of villages until 360 participants have been enrolled. The investigators expect enrolment from approximately 10 villages.

A trained, Khmer-speaking enumerator will conduct an interview in the participants home. The questionnaire will collect demographic data, as well as information on dietary intake (including fish sauce), thoughts and perceptions of fortified products, and knowledge of thiamin deficiency and beriberi. Once the questionnaire is complete the participant will walk with the interviewer to a central meeting spot within the village (typically the Village Chief's home) to complete anthropometric measurements (height and weight). The next morning the participant will travel to the local health centre for a non-fasted blood draw.

Once the participant completes the baseline questionnaire, anthropometrics, and blood collection she will be randomly assigned to one of the three treatment groups: low concentration thiamin-iron-fortified fish sauce (2mg thiamin/mL fish sauce + iron), higher concentration thiamin-fortified fish sauce (8mg thiamin/mL fish sauce + iron), or placebo: iron-fortified fish sauce. The bottles and labels of the three fish sauces will be identical in appearance, except for a code that differentiates the sauces.

All participants will be visited biweekly for monitoring and evaluation of fish sauce consumption. Fish sauce will be distributed during these visits to ensure that there are no 'stock outs' of fish sauce during the study.

Within the first month of the study all participants will attend an educational workshop with training regarding dietary thiamin intake, thiamin deficiency and beriberi, and infant and young child feeding (IYCF) practices.

Anthropometric measurements (weight and length) will be taken within 72 hours of the birth of the participant's infant (t~3 months).

At t~4 months, a subset of households (n=28) will participate in an Observed Weighed Fish Sauce Record wherein a trained enumerator measure all fish sauce consumed by the participant throughout one day. Two repeat observed weighed fish sauce records will be completed within a 2 week period.

At endline (t=6 months), the questionnaire, anthropometrics, and blood draw will be repeated with all women. The investigators will also collect a venous blood sample (4mL) from the infant, and a breast milk sample from mothers from the pregnant cohort. Investigators plan to analyze all samples within two months of the endline sample collection, and will return to the villages to share study findings with all participants at a community meeting (general results shared), and then separately to share individual thiamin results one-on-one. All participants will have already participated in an educational workshop highlighting the importance of dietary thiamin intake, and the signs of thiamin deficiency and beriberi. Individuals with suboptimal thiamin status will be encouraged to speak with their healthcare provider, and will also be counselled using the materials that were previously used in the educational workshop.

ELIGIBILITY:
Inclusion Criteria:

Women of Childbearing Age Cohort:

* be the female head of their household,
* have at least one child between 12 - 59 months of age at baseline,
* be living in Prey Veng province, Cambodia, and not planning to move in the next six months,
* agree to exclusively feed her entire household the study fish sauce for six months, and
* be willing to provide venous blood samples at baseline and endline.

Pregnant Women Cohort:

* be the female head of their household,
* be ~3-8 mo pregnant with a singleton fetus at baseline,
* have no prior history of preeclampsia, pre-term delivery, or birth defects,
* know her approximate due date,
* be living in Prey Veng province, Cambodia, and not planning to move in the next six months,
* agree to exclusively feed her entire household the study fish sauce for six months, and
* be willing to provide venous blood samples at baseline and endline, a breast milk sample at endline, and to allow for a blood sample to be taken from her infant (aged ~3 months) at endline.

Exclusion Criteria:

Women of Childbearing Age Cohort:

* not be receiving any other intervention (for example, homestead food production),
* not be pregnant or hoping to become pregnant within the next 6 months, and
* not be taking any supplement that contains thiamin.

Pregnant Women Cohort:

* not be receiving any other intervention (for example, homestead food production), and
* not be taking any supplement that contains thiamin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Erythrocyte thiamin diphosphate | Baseline (t=0), Endline (t=6 months)
  Measurement at baseline and endline for all women. Blood samples from infants of women recruited in the pregnancy cohort will be collected at endline only.

SECONDARY OUTCOMES:
Breast milk thiamin concentration | Endline (t=6 months)
  Breast milk will collected only from those women recruited in the pregnancy cohort (n=90)

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Green, PhD, Principal Investigator — University of British Columbia; Kyly C Whitfield, MSc, Study Director — University of British Columbia; Judy McLean, PhD, Study Chair — University of British Columbia; Zaman Talukder, MPH, Study Chair — Helen Keller International
Locations (1):
- (Various Villages), Prey Veng, Cambodia

REFERENCES:
- [Derived] Whitfield KC, Karakochuk CD, Kroeun H, Sokhoing L, Chan BB, Borath M, Sophonneary P, Moore K, Tong JKT, McLean J, Talukder A, Lynd LD, Li-Chan ECY, Kitts DD, Green TJ. Household Consumption of Thiamin-Fortified Fish Sauce Increases Erythrocyte Thiamin Concentrations among Rural Cambodian Women and Their Children Younger Than 5 Years of Age: A Randomized Controlled Efficacy Trial. J Pediatr. 2017 Feb;181:242-247.e2. doi: 10.1016/j.jpeds.2016.10.066. Epub 2016 Dec 7. PMID 27939124
- [Derived] Whitfield KC, Karakochuk CD, Kroeun H, Hampel D, Sokhoing L, Chan BB, Borath M, Sophonneary P, McLean J, Talukder A, Lynd LD, Li-Chan EC, Kitts DD, Allen LH, Green TJ. Perinatal Consumption of Thiamine-Fortified Fish Sauce in Rural Cambodia: A Randomized Clinical Trial. JAMA Pediatr. 2016 Oct 3;170(10):e162065. doi: 10.1001/jamapediatrics.2016.2065. Epub 2016 Oct 3. PMID 27532780